CLINICAL TRIAL: NCT03249961
Title: How Many Days Would You Want to Practice a Skill to Achieve it?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 175-2017
Record Dates: First submitted 2017-08-02; First posted 2017-08-15 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Motor Learning
Keywords: motor; transcranial direct current stimulation; transcranial magnetic stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Brain stimulation (Experimental): Participants will receive Sham TDCS, and Transcranial Magnetic Stimulation (TMS)
  Interventions: Device: Sham TDCS; Device: Transcranial Magnetic Stimulation (TMS)
- Excitatory Brain Stimulation (Experimental): Participants will receive Anodal TDCS, and Transcranial Magnetic Stimulation (TMS)
  Interventions: Device: Anodal TDCS; Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Sham TDCS — Placebo stimulation is applied to the left motor cortex while participants perform a motor task in the right hand. During the motor task, participants use their right hand to pinch a force transducer that controls an on-screen cursor to navigate between a start position and a sequence of 5 other positions to the right.
  Arms: Placebo Brain stimulation
Device: Anodal TDCS — Excitatory stimulation is applied to the left motor cortex while participants perform a motor task in the right hand. During the motor task, participants use their right hand to pinch a force transducer that controls an on-screen cursor to navigate between a start position and a sequence of 5 other positions to the right.
  Arms: Excitatory Brain Stimulation
Device: Transcranial Magnetic Stimulation (TMS) — Participants will receive Transcranial Magnetic Stimulation (TMS) to allow research investigators to determine the location of the left motor cortex.

SUMMARY:
Practice is required to improve your shot in basketball or to play a musical instrument. The learning of these motor skills can be further enhanced by non-invasively stimulating regions of the brain that control movements with electrical currents. These electric currents can strengthen or weaken connections of the brain, which consequently affects a person's ability to improve their performance on a skill. Non-invasive brain stimulation (NIBS) is widely applied in many disciplines of neuroscience research, and has potential therapeutic application. There are two specific types of NIBS that will be used in this research study: 1) Transcranial Direct Current Stimulation (tDCS), which applies very weak electrical currents via two rubber electrodes on the scalp, and 2) Transcranial Magnetic Stimulation (TMS), which applies magnetic pulses via a coil against the head, to stimulate regions of the brain. Both types of non-invasive brain stimulation (i.e., tDCS, and TMS) are well-tolerated, painless, and safe. The application of tDCS to brain regions that control movements, concurrently with practice of a skill, results in better skill performance, than practice alone with no tDCS. Therefore, in this study, we will be testing different types of brain stimulation and different amounts of practice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* prior history of neurological or psychiatric disease
* prior experience with the motor task used
* contraindications to TMS and TDCS (e.g., metal implants, history of seizures and headaches)
* musculoskeletal injury to upper limb
* drugs that interact with NIBS (e.g., antidepressants, antipsychotics, anticonvulsants)

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Accuracy | Up to 8 days
  Accuracy is defined as the proportion of trials per block with hits to all targets in the correct sequence order.
Speed | Up to 8 days
  Speed is captured by the average sequence movement time per training block

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chen, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada